CLINICAL TRIAL: NCT03373695
Title: A Multicenter, Randomized, Controlled Clinical Study to Evaluate the Efficacy and Safety of Dissolve™ Compared to SeQuent® Please in Treatment of Coronary In-stent Restenosis in Chinese Population
Brief Title: A Safety and Efficacy Study of Dissolve™ in Treatment of Coronary In-stent Restenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DK Medical Technology (Suzhou) Co., Ltd. (Industry)
Collaborators: Core Medical (Beijing) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-VP-01
Record Dates: First submitted 2017-12-05; First posted 2017-12-14 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Coronary In-stent Restenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dissolve™ (Experimental)
  Interventions: Device: Dissolve™
- SeQuent®Please (Active Comparator)
  Interventions: Device: SeQuent®Please

INTERVENTIONS:
Device: Dissolve™ — Dissolve™ are to be used in the trial
  Arms: Dissolve™
Device: SeQuent®Please — SeQuent®Please are to be used in the trial
  Arms: SeQuent®Please

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of treatment of coronary in-stent restenosis by Paclitaxel-eluting balloon catheter Dissolve™ versus SeQuent®Please, and the reference diameter of coronary artery stenosis is 2.5mm-4.0mm and the length ≤ 26mm.

ELIGIBILITY:
Inclusion Criteria:

Related to the patients:

1. Age ≥18 years old
2. Patients who agree to accept the angiography follow-up visit at 9-month and follow up visits at 1-month, 6-month, 9-month, 1-year, 2-year, 3-year, 4-year and 5-year
3. Patients with stable angina, unstable angina, old myocardial infarction or proven asymptomatic ischemia
4. Patients who can receive any kind of coronary revascularization (including balloon angioplasty, stent implantation or coronary artery bypass grafting)

   Related to lesion:
5. Restenosis after the first stent implant (including bare metal stents, stents with inert coating, and stents with active coating): Type Mehran I, Type II and Type III; the reference blood vessel diameter is 2.5 mm-4.0 mm, length ≤ 26mm
6. Before surgery, stenosis diameter must be ≥ 70% or ≥ 50% and accompanied by ischemia
7. The distance between other lesion requires interventional therapy and the target lesion must be > 10mm
8. One subject is allowed to have 2 target lesions at most, and 1 paclitaxel drug balloon for each lesion for dilation
9. Residual stenosis must be ≤ 30% after pre-dilatation, and dissection must be ≤ NHLBI type B

Exclusion Criteria:

Related to patients

1. Pregnant or lactating women, or women who plan to get pregnant within 12 months or refuse to take effective contraceptives
2. Patients with cardiogenic shock
3. The patients had cerebral stroke within 6 months before being included, or have a history of peptic ulcer or gastrointestinal bleeding, or the patients have a bleeding tendency according to the investigator. Patients who are forbidden to use anticoagulation agents or anti-platelet drugs, and unable to tolerate aspirin or clopidogrel. Patients who are not able to tolerate and comply with dual antiplatelet therapy for at least 3 months after operation
4. Patients who have Myocardial Infarction with thrombus or coronary slow flow symptoms and require immediate intervention
5. Patients who had ST-Elevation Myocardial Infarction within 1 week before being included
6. Patients with severe congestive heart failure or NYHA grade IV heart failure
7. Patients with moderate or severe valvular heart disease
8. Patients who had heart transplantation
9. Patients with renal insufficiency (eGFR < 30mL/min)
10. The patients have a life expectancy of less than 12 months, or it would be difficult to finish follow-ups within 12 months.
11. The patients are participating in any other clinical trials before reaching the primary endpoints
12. Patients who are unsuitable for the study according to the investigator due to other reasons

    Related to the Lesion:
13. Patients with total occlusion at the target lesion
14. Lesion which cannot be treated by percutaneous transluminal coronary angioplasty (PTCA) or percutaneous intervention (PCI)
15. Reference vessel diameter < 2.0mm
16. Patients with multiple lesions (≥ 3) requiring percutaneous coronary intervention treatment in the same artery
17. 3-vessel disease that all need to be intervened
18. The diameter of the branch lesions in the target lesion ≥ 2.5mm
19. LM lesions and Ostial lesion within 5mm to the root aorta
20. Non-target lesion was not intervened successfully before target lesions being intervened

    Related to concomitant therapy:
21. Patients cannot tolerate aspirin and/or clopidogrel and or tricagrelor, patients with the history of neutrocytopenia or thrombocytopenia, or patients with severe hypohepatia and prohibited to take clopidogrel
22. Patients known allergic to paclitaxel
23. Patients known allergic to contrast materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
In-segment Late Lumen Loss | From the end of procedure to 9 months after the procedure
  In-segment late lumen loss is defined as the change in minimal lumen diameter (MLD) within the margins of the device and 5 mm proximal and 5 mm distal to the device from post-procedure to 9 months by angiography.

SECONDARY OUTCOMES:
Device success rate of the interventional therapy | From the start of index procedure to end of index procedure
  Successful delivery and use of the assigned balloon at the intended target lesion and successful withdrawal of the delivery system with attainment of final residual stenosis of less than 30% and TIMI 3 blood flow by visual estimation.
Lesion success rate of the interventional therapy | From the start of index procedure to end of index procedure
  Attainment of final residual stenosis of target lesion less than 30% and TIMI 3 blood flow by visual estimation.
Clinical success rate of the interventional therapy | 7 days after the procedure
  Achievement of final residual stenosis of less than 30% by visual estimation with successful delivery and use of assigned balloon at the intended target lesion and successful withdrawal of the delivery system for the target lesion without the occurrence of cardiac death, target vessel Myocardial Infarction (MI) or repeat Target lesion revascularization (TLR).
Rate of restenosis in the target lesions | 9 months after the procedure
  Restenosis is defined as stenosis > 30% by angiography
TLR rate | 9 months after the procedure
Target vessel revascularization (TVR) rate | 9 months after the procedure
Target lesion failure (TLF) rate | 9 months after the procedure
Rate of major adverse cardiovascular events | 1 month, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years after the procedure
Rate of all adverse events and severe adverse events | 1 month, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Shubin Qiao, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (15):
- China (15):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University People's Hospital, Capital Medical University, Beijing
  - Xiangya Hospital of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - The Second Affiliated Hospital of Dalian Medical University, Dalian
  - General Hospital of Daqing Oil Field, Daqing
  - Sir Run Run Shaw Hospital, Zhejiang University School of medicine, Hangzhou
  - The First Affiliated Hospital of Zhengzhou University, Hangzhou
  - Union Hospital, Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - General Hospital of Ningxia Medical University, Yinchuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu S, Zhou Y, Shen Z, Chen H, Qiu C, Fu G, Li H, Yu Z, Zeng Q, Li Z, Li W, Qiao S; Dissolve ISR Investigators. A Randomized Comparison of 2 Different Drug-Coated Balloons for In-Stent Restenosis. JACC Cardiovasc Interv. 2023 Apr 10;16(7):759-767. doi: 10.1016/j.jcin.2022.12.018. PMID 37045496